CLINICAL TRIAL: NCT06669650
Title: Personalized Post-Operative Opiate Prescriptions Based on Pharmacogenetics of CytochromeP450, COMT, and OPRM1
Brief Title: Personalized Post-Operative Pain Management
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Trey Henderson, Study Coordinator, University of Tennessee Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5226; CORNET Award (Other Grant/Funding Number: The University of Tennessee Graduate School of Medicine)
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Persistent Post Operative Opioid Use; Post-surgical Pain
Keywords: CYP2D6 SNPs; OPRM1 SNPs; COMT SNPs; Pharmacogenomics
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone; Hydromorphone

STUDY DESIGN:
Intervention Model Description: Standard of Care (oxycodone) versus intervention group (hydromorphone)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard post-operative pain management (control) (Active Comparator): Patients in the control groups will follow the current hospital standard of care and receive oxycodone 5mg every 4 hours as needed for moderate pain and oxycodone 10mg every four hours as needed for severe pain.
  Interventions: Other: PGx guided personalized post-operative pain management; Drug: Oxycodone
- Pharmacogenomics (PGx) guided treatment (hydromorphone) (Experimental): Patients who are poor CYP2D6 metabolizers or rapid CYP2D6 metabolizers with moderate or severe pain, will be prescribed either oral hydromorphone 2mg every 4 hours as needed or oral hydromorphone 4mg every 4 hours as needed, respectively.
  Interventions: Other: PGx guided personalized post-operative pain management; Drug: Hydromorphone

INTERVENTIONS:
Other: PGx guided personalized post-operative pain management — Patients in the intervention group will receive post operative opioid therapy based on their pharmacogenomic results. Patients who are poor CYP2D6 metabolizers or rapid CYP2D6 metabolizers with moderate or severe pain, will be prescribed either oral hydromorphone 2mg every 4 hours as needed or oral hydromorphone 4mg every 4 hours as needed, respectively. Patients who are intermediate or normal CYP2D6 metabolizers with moderate or severe pain will receive oxycodone 5mg or oxycodone 10mg every 4 hours as needed respectively similar to the treatment offered to the control subjects. Normal or intermediate CYP2D6 metabolizers who are concomitantly taking a drug which is a strong CYP2D6 inducer will be treated as if they are in the rapid metabolizer group, and normal or intermediate patients that are concomitantly taking a drug which is a strong CYP2D6 inhibitor will be treated as if they were a poor metabolizer.
Drug: Oxycodone — oxycodone
  Arms: Standard post-operative pain management (control)
Drug: Hydromorphone — hydromorphone
  Arms: Pharmacogenomics (PGx) guided treatment (hydromorphone)

SUMMARY:
The main questions this study aims to answer are:

Does perioperative PGx personalized opiate therapy reduce persistent post-operative opioid use dependency, improve pain management and reduce opiate related adverse events in opioid naïve patients after surgery?

Participants will:

Take hydromorphone if the PGx results determine they have a SNP indicating high or low metabolic activity in the CYP2D6 enzyme.

Complete a 7-day pain diary post-discharge. Complete a follow-up phone call once per month for 90 days.

ELIGIBILITY:
Inclusion Criteria:

1.18-85 years of age 2.Able to read and understand study procedures. 3.Willing to participate and sign an ICF. 4.Opioid naïve 90 days prior to surgery.

Exclusion Criteria:

1. <18 years of age and >85 years of age
2. Unable to understand study procedures.
3. Unwilling to give consent.
4. Patients with cognitive impairment that can affect their ability to give consent.
5. Previous Surgery <14 days from time of enrollment.
6. Allergies to study intervention or oxycodone.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Persistent Post-Operative Opioid Use | 90 days
  To determine the overall difference in the number of post-operative opioid prescriptions in 90 days using PGx guided post operative medication

SECONDARY OUTCOMES:
Post-Surgical Pain | 7 days
  To determine if PGx guided medication improves post-operative pain scores compared to similar patients who are given the standard current post operative opiate treatment. The scores are being rated using the Face, Legs, Activity, Cry and Consolability scale ranging from a minimum value of 0 to a maximum value of 10.

OTHER OUTCOMES:
Opioid Related Adverse Events | 90 days
  To determine if PGx guided medication reduces total opioid related adverse events compared to standard post operative opiate therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Tennessee Graduate School of Medicine, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided